CLINICAL TRIAL: NCT04942535
Title: STEP Together: A Hybrid Type 1 Effectiveness-Implementation Study of Social Incentives Strategies to Increase Physical Activity
Brief Title: STEP Together: An Effectiveness-Implementation Study of Social Incentives and Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 02022; 1R01HL152430 (NIH); 842677 (Other: IRB Number)
Record Dates: First submitted 2021-06-17; First posted 2021-06-28 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Physical Activity
Keywords: Physical Activity; Older Adults; Gamification; Social Incentives; Charity; Family
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Social Incentive Gamification (Experimental): Each participant is enrolled as part of a family team. Each participant wears a Fitbit every day and strives to achieve their daily step goal.
  Participants in this arm receive the Social Incentive Gamification intervention during the 12 month intervention and Daily Performance Feedback during the 6 month follow up.
  Interventions: Behavioral: Social Incentive Gamification; Behavioral: Daily Performance Feedback
- Social Goals through Incentives to Charity (Experimental): Each participant is enrolled as part of a family team. Each participant wears a Fitbit every day and strives to achieve their daily step goal.
  Participants in this arm receive the Social Goals through Incentives to Charity intervention during the 12 month intervention and Daily Performance Feedback during the 6 month follow up.
  Interventions: Behavioral: Social Goals through Incentives to Charity; Behavioral: Daily Performance Feedback
- Control (Active Comparator): Each participant is enrolled as part of a family team. Each participant wears a Fitbit every day and strives to achieve their daily step goal.
  Participants in this arm receive Daily Performance Feedback during the 12 month intervention and 6 month follow up.
  Interventions: Behavioral: Daily Performance Feedback

INTERVENTIONS:
Behavioral: Social Incentive Gamification — Participants enroll as a family team. They are asked to use a Fitbit activity tracker daily. Each participant sets a daily step goal based on their baseline step count.
  Each participant signs a pre-commitment contract. Participants are entered into a game with their family members. Each family receives 70 points weekly. Each day, a family member is selected at random to represent the family. If that person's step goal was achieved, the family keeps its points; if not, they lose 10 points. The participant is notified the following day if they were the family rep.
  At the end of the week, if the family has 40 points or more, they advance 1 level. If they have less than 40 points, the family drops down 1 level. Each family team starts in the middle of 5 levels.
  At the end of the intervention, families in the top 2 levels receive a small gift.
  In the 6 month follow-up, participants receive a daily text message stating whether or not they achieved their step goal on the prior day.
  Arms: Social Incentive Gamification
Behavioral: Social Goals through Incentives to Charity — Participants enroll as a family team. They are asked to use a Fitbit activity tracker daily. Each participant sets a daily step goal based on their baseline step count.
  Families select a charity at the beginning of the intervention. They are informed that $20 is available each week to be donated to a charity of their choice. Each day, a family member is selected at random to represent the family. If that person's step goal was achieved, the family gets credit for meeting their goal; if not, the entire family does not get credit. The participant is notified the following day if they were the family rep.
  If the family achieves their goal on at least 4 of 7 days in a week, $20 is donated to charity.
  In the 6 month follow-up, participants receive a daily text message stating whether or not they achieved their step goal on the prior day.
  Arms: Social Goals through Incentives to Charity
Behavioral: Daily Performance Feedback — Participants enroll as a family team. They are asked to use a Fitbit activity tracker daily. Each participant sets a daily step goal based on their baseline step count.
  Participants receive a daily text message stating whether or not they achieved their step goal on the prior day.

SUMMARY:
Higher levels of physical activity have been demonstrated to improve health across a wide range of contexts and reduce cognitive decline as adults become older, but more than half of all adults in the United States do not meet their physical activity goals. One type of physical activity that is broadly applicable to people of all ages is walking. This study will use a Hybrid Type 1 effectiveness-implementation design to adapt and test the effectiveness of two successful social incentive-based interventions, a gamification strategy and financial incentives donated to charity on the participants behalf, to increase physical activity among low-income, mostly minority families in community settings.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and speak English;
* Has a smartphone or tablet;
* Lives in the Philadelphia area;
* Age 14 or older;
* Able to provide informed consent;
* Enrolled as a member of a 2 to 10 member family team with least one member 60 years or older.

Exclusion Criteria:

* Already participating in another physical activity study;
* An 18-month physical activity program is infeasible (e.g., metastatic cancer, unable to ambulate or provide informed consent) or unsafe (currently pregnant or told by a physician not to exercise);
* Do not have sufficient eyesight or dexterity to operate device;
* Average step count greater than 7,500 steps/day during the run-in period.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 779 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-10-11 (Actual)

PRIMARY OUTCOMES:
Change in mean daily step counts during the 12 month intervention | Months 1-12
  Change in mean daily steps from baseline to the end of the 12 month intervention period. Steps will be measured using the Fitbit Inspire 2 wearable device.

SECONDARY OUTCOMES:
Change in mean daily step counts during the 12 month intervention and 6 month follow up | Months 1-18
  Change in mean daily steps from baseline to the end of the 12 month intervention and 6 month follow up. Steps will be measured using the Fitbit Inspire 2 wearable device.
Change in mean minutes of moderate-to-vigorous physical activity (MVPA) during the 12 month intervention | Months 1-12
  Change in mean daily minutes of MVPA from baseline to the end of the 12 month intervention period. Minutes of MVPA will be measured using the Fitbit Inspire 2 wearable device.
Change in mean minutes of moderate-to-vigorous physical activity (MVPA) during the 12 month intervention and 6 month follow up | Months 1-18
  Change in mean daily minutes of MVPA from baseline to the end of the 12 month intervention and 6 month follow up. Minutes of MVPA will be measured using the Fitbit Inspire 2 wearable device.
Difference in proportion of weeks physical activity guidelines were achieved during the 12 month intervention | Months 1-12
  Difference between study arms in the proportion of weeks that physical activity guidelines (150 minutes per week of MVPA) were achieved. Minutes of MVPA will be measured using the Fitbit Inspire 2 wearable device.
Difference in proportion of weeks physical activity guidelines were achieved during the 12 month intervention and 6 month follow up | Months 1-18
  Difference between study arms in the proportion of weeks that physical activity guidelines (150 minutes per week of MVPA) were achieved. Minutes of MVPA will be measured using the Fitbit Inspire 2 wearable device.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Glanz, PhD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available.

REFERENCES:
- [Derived] Scheffey K, Aronson J, Goncalves Y, Greysen SR, Iwu A, Kwong PL, Nezir F, Small D, Glanz K. Design and baseline characteristics of an implementation study to increase activity with social incentives: The STEP together trial. Contemp Clin Trials. 2025 Jun;153:107909. doi: 10.1016/j.cct.2025.107909. Epub 2025 Apr 10. PMID 40216076

DOCUMENTS (1):
  • Informed Consent Form (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/35/NCT04942535/ICF_000.pdf